CLINICAL TRIAL: NCT06234137
Title: A Prospective, Open, Multicenter Single-arm Clinical Studie of Docetaxel, Carboplatin Combined With Inetetamab and Pyrotinib in the Treatment of Local-advanced HER2-positive Breast Cancer
Acronym: neoPICD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wang Ouchen (Other)
Responsible Party: Sponsor-Investigator, Wang Ouchen, Chief Physician, First Affiliated Hospital of Wenzhou Medical University
Organization: First Affiliated Hospital of Wenzhou Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2021-113
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Breast Neoplasm Female
MeSH Terms: interventions — Docetaxel; Carboplatin; pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental)
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Drug: Inetetamab; Drug: Pyrotinib

INTERVENTIONS:
Drug: Docetaxel — 75mg/m2 iv escalating to 100mg/m2 iv 3-weekly
Drug: Carboplatin — AUC=6 min/mL iv 3-weekly
Drug: Inetetamab — 8mg/kg iv loading dose, followed by 6mg/kg iv 3-weekly
  Other Names: cipterbin
Drug: Pyrotinib — 400mg orally daily

SUMMARY:
This study is a prospective, open, multi-center, single arm trial. The treatment group will receive six cycles of docetaxel, carboplatin combined with Inetetamab and Pyrotinib before surgery. By focusing on tpCR (ypT0/is, ypN0) evaluated by pathology, the efficacy of docetaxel, carboplatin combined with Inetetamab and Pyrotinib in the preoperative treatment of locally advanced HER2-positive breast cancer will be evaluated. During long-term follow-up, event-free survival (EFS), disease-free survival (DFS), distant metastasis-free survival (DDFS), overall survival (OS), central nervous system disease-free survival (CNSDFS) under this treatment regimen will be evaluated, and the efficacy-related biomarkers will be explored. The cardiotoxicity of Inetetamab and Pyrotinib in the treatment of breast cancer is also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-75 years old;
2. ECOG score 0-1;
3. Breast cancer meets the following criteria: Histologically confirmed invasive breast cancer, primary tumor diameter > 2 cm as determined by standard evaluation methods at the research center; tumor stage: locally advanced;
4. HER2 expression-positive breast cancer confirmed by pathological examination;
5. Known hormone receptor status (ER and PR);
6. The functional level of major organs must meet the following requirements (no blood transfusion within 2 weeks before screening, no use of white blood cell and platelet-raising drugs):

(1) Blood routine: neutrophil (ANC) >= 1.5×10^9/L; platelet count (PLT) >= 90×10^9/L; hemoglobin (Hb) >= 90 g/L; (2) Blood biochemistry: total bilirubin (TBIL) <= upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 1.5×ULN; alkaline phosphatase <= 2.5×ULN; urea nitrogen (BUN) and creatinine (Cr) <= 1.5×ULN; (3) Echocardiography: left ventricular ejection fraction (LVEF) >= 60%; (4) 12-lead ECG: Fridericia-corrected QT interval (QTcF) < 470 msec; 7. Female patients who are not menopausal or surgically sterilized: agree to abstain from sex or use effective contraceptive methods during treatment and for at least 7 months after the last dose in the study treatment; 8. Voluntarily join the study, sign the informed consent, have good compliance and are willing to cooperate with follow-up.

Exclusion Criteria:

1. IV (metastatic) breast cancer;
2. Received anti-tumor therapy or radiotherapy for any malignant tumor in the past, excluding cured cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma and other malignant tumors;
3. Receiving anti-tumor therapy in other clinical trials at the same time, including endocrine therapy, bisphosphonate therapy or immunotherapy;
4. Received major surgical operations unrelated to breast cancer within 4 weeks before enrollment, or the patient has not fully recovered from such surgical operations;
5. Severe cardiac disease or discomfort, including but not limited to the following: a history of heart failure or systolic dysfunction (LVEF < 60%); high-risk uncontrolled arrhythmias, such as atrial tachycardia, resting heart rate > 100 bpm , significant ventricular arrhythmia (eg, ventricular tachycardia) or higher-grade AV block (ie, Mobitz II second-degree AV block or third-degree AV block); antianginal medication indicated angina pectoris; clinically significant heart valve disease; transmural myocardial infarction on ECG; poorly controlled hypertension (systolic > 180 mmHg and/or diastolic > 100 mmHg);
6. Inability to swallow, intestinal obstruction, or other factors that affect drug taking and absorption;
7. Those who are known to have a history of allergy to the drug components of this regimen; have a history of immunodeficiency, including HIV positive test, or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;
8. Female patients during pregnancy and lactation, female patients with fertility and positive baseline pregnancy test, or patients of childbearing age who are unwilling to take effective contraceptive measures during the entire trial period and within 7 months after the last study drug;
9. Have serious comorbidities or other comorbidities that would interfere with planned treatment, or any other condition that the investigator considers the patient unsuitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2021-11-27 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
tpCR | Approximately 5 months from randomization following surgery or early withdrawal, whichever occurred first (Surgery was performed within 2 weeks after Cycle 6)
  total pathological complete response

SECONDARY OUTCOMES:
EFS | Randomization up to a maximum of 329 weeks
  Event-free survival
DFS | Randomization up to a maximum of 329 weeks
  Disease-free survival
DDFS | Randomization up to a maximum of 329 weeks
  Distant disease free survival
OS | Up to 2 years
  Overall survival
CNS-DFS | Randomization up to a maximum of 329 weeks
  Central nervous system disease-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China